CLINICAL TRIAL: NCT03472417
Title: Partial Rebreathing in the Treatment of Migraine With Aura
Acronym: CapnoMigra
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Rehaler (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2016-003683-39
Record Dates: First submitted 2017-05-02; First posted 2018-03-21 (Actual); Last update posted 2018-03-23 (Actual); Status verified 2016-11

CONDITIONS: Migraine With Aura
MeSH Terms: conditions — Migraine with Aura

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active partial rebreathing device (Active Comparator)
  Interventions: Device: Active partial rebreathing device
- Dummy partial rebreathing device (Sham Comparator)
  Interventions: Device: Dummy partial rebreathing device

INTERVENTIONS:
Device: Active partial rebreathing device
  Arms: Active partial rebreathing device
Device: Dummy partial rebreathing device
  Arms: Dummy partial rebreathing device

SUMMARY:
A study to test the efficacy of a partial rebreathing device in treating and/or preventing migraine pain

ELIGIBILITY:
Inclusion Criteria:

* - Migraine with aura
* Attack frequency of between one and six migraine-with-aura attacks per month over the last six months
* Adults (18-60 years)
* Age at onset of migraine < 50 years
* If taking migraine prophylactic drugs, the dosis must have been stable for > 3 months
* Must speak and understand Danish

Exclusion Criteria:

* - Cardiovascular disease, pulmonary disease, metabolic acid/base disorder, cancer, moderate and severe depression, anemia or other blood disease
* Chronic migraine, i.e. more than 15 headache days per month over the last three months
* Medication overuse headache
* More than six migraine-with-aura attacks per month
* Non-migraine headache on more than six days per month
* A typical duration between migraine-with-aura attacks of less than 48 hours

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2016-11; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Headache Intensity Difference at 0 vs 2 hours post-treatment | 2 hours
  0-3 point scale (0 = none, 1 = mild, 2= moderate, 3 =severe)

SECONDARY OUTCOMES:
Headache Intensity Difference at 0 and 1 hour post-treatment (0-3 point scale) | 1 hour
  0-3 point scale (0 = none, 1 = mild, 2= moderate, 3 =severe)
Pain reduction/relief at 1 hour | 1 hour
  percentage of study participants reporting no or mild pain 1 hour after first using the device
Pain reduction/relief at 2 hours | 2 hours
  percentage of study participants reporting no or mild pain 2 hours after first using the device
Nausea Intensity Difference 0 vs 1 hour post-treatment | 1 hour
  0-3 scale (0 = none, 1 = mild, 2= moderate, 3 =severe)
Nausea Intensity Difference 0 vs 2 hours post-treatment | 2 hours
  0-3 scale (0 = none, 1 = mild, 2= moderate, 3 =severe)
Photo - and/or phono-phobia Intensity Difference 0 vs 1 hour post-treatment | 1 hour
  0-3 scale (0 = none, 1 = mild, 2= moderate, 3 =severe)
Photo - and/or phono-phobia Intensity Difference 0 vs 2 hours post-treatment | 2 hours
  0-3 scale (0 = none, 1 = mild, 2= moderate, 3 =severe)
Functional Disability Difference 0 vs 1 hour post-treatment | 1 hour
  0-3 scale (0 = none, 1 = mild, 2= moderate, 3 =severe)
Functional Disability Difference 0 vs 2 hours post-treatment | 2 hours
  0-3 scale (0 = none, 1 = mild, 2= moderate, 3 =severe)
Sustained pain freedom at 24 hours | 24 hours
  percentage of study participants who are pain free 24 hours after device use
Treatment preference vs. patient's normal treatment | 24 hours
  -2 to +2 scale ((-2 = much worse than normal treatment, - 1 = somewhat worse, 0 = no difference, +1 = somewhat better, +2 = much better))
Aura symptoms aborted after one use of device | 20 minutes
  yes/no
Side effects | through study completion (1 to 10 months)
  Qualitative analysis
Adverse events | through study completion (1 to 10 months)
  Qualitative analysis
Medicine use in 24 hours after device use | 24 hours
  qualitative comparison

CONTACTS AND LOCATIONS:
Overall Officials: Flemming W Bach, MD, PhD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Pain and Headache Clinic, Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fuglsang CH, Johansen T, Kaila K, Kasch H, Bach FW. Treatment of acute migraine by a partial rebreathing device: A randomized controlled pilot study. Cephalalgia. 2018 Sep;38(10):1632-1643. doi: 10.1177/0333102418797285. Epub 2018 Aug 22. PMID 30134739